CLINICAL TRIAL: NCT03844698
Title: Outcome Study of Sarcoidosis: a New Paraneoplastic Syndrome in Patient With Cancer
Brief Title: Association Between Cancer and Sarcoidosis
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Other Study IDs: 20180852
Record Dates: First submitted 2019-02-11; First posted 2019-02-18 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Sarcoidosis; Cancer
Keywords: sarcoidosis, cancer, paraneoplastic, treatment, outcome
MeSH Terms: conditions — Sarcoidosis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Pathological slides from patients, which contains Hematoxylin and Eosin ( H&E) tissue stain fixation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Sarcoidosis and Cancer: These group of patients have a diagnosis of Sarcoidosis and Cancer on the Pathological Report.

SUMMARY:
The purpose of this study is to develop a clinical dataset of sarcoidosis patients with a diagnosis of cancer who are categorized by date of birth, sex, race/ethnicity, clinical information, laboratory and imaging information, time of sarcoidosis onset, cancer type and treatment, time of cancer diagnosis, stage and grade.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Sarcoidosis following cancer
* Granulomatous reaction must be proven by pathology

Exclusion Criteria:

. Aged younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer who were seeking or receiving medical care at the University of Miami that satisfy the inclusion and exclusion criteria of study are eligible to participate.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Pathology Proven Sarcoidosis In Patients with Cancer | up to 10 years
  Number of Participants With Sarcoidosis Events as Assessed by Positive Granulomatous Reaction in the Biopsies of Lung, Mediastinal Lymph Nodes, or Other Organs After Cancer Diagnosis.

SECONDARY OUTCOMES:
Cancer Cytogenetics and Sarcoidosis | up to 10 years
  Number of Participants With Sarcoidosis Events as Assessed by Cancer Cytogenetic Profiles of Cancer.
Treatment Requirement of Sarcoidosis | up to 10 years
  Number of Participants With Sarcoidosis Events as Assessed by Requirement of Treatment with Steroid or Other Anti-Sarcoid Medications in Patients with Cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Mirsaeidi, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murthi M, Yoshioka K, Cho JH, Arias S, Danna E, Zaw M, Holt G, Tatsumi K, Kawasaki T, Mirsaeidi M. Presence of concurrent sarcoid-like granulomas indicates better survival in cancer patients: a retrospective cohort study. ERJ Open Res. 2020 Oct 26;6(4):00061-2020. doi: 10.1183/23120541.00061-2020. eCollection 2020 Oct. PMID 33263026